CLINICAL TRIAL: NCT06909526
Title: Implementation of a Short Mindfulness-based Program for Young Women in Puerto
Brief Title: Implementation of a Short Mindfulness-based Program for Young Women in Puerto Rico
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Andrea Lopez-Cepero, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00007906
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Stress; Anxiety
Keywords: Stress in women; Anxiety in women; Mindfullness; Mindfulness-based stress reduction
MeSH Terms: conditions — Anxiety Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBSR: Mindfulness-based stress reduction (Experimental): * 4-week intervention (1 weekly virtual session; daily mindfulness exercises at home)
  * 3 study assessments (baseline, post-intervention, 1 month post-intervention)
  Interventions: Behavioral: Mindfulness-based stress reduction :MBSR
- Usual care group (Placebo Comparator): Placebo Comparator: Usual care group
  * No intervention, but participants will have access to audio files and a mindfulness information sheet after study completion
  * 3 study assessments (baseline, 1 mo, 2mo)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction :MBSR — The intervention consists of 4 weekly virtual sessions and daily mindfulness exercises at home (between 1-5min of duration each, according to the participant's availability. Each session lasts 1 hour (except the first one, which is 1.5 hours due to discussion of the program's logistics). The sessions follow a brief check-in, a lecture on the week's topic, and a guided practice exercise. For the audio guides, participants can select a short version of the daily practice exercise or a longer one, which they will record in the practice logs. Participants also receive information sheets summarizing the weekly sessions.
  Other Names: MBSR
  Arms: MBSR: Mindfulness-based stress reduction
Behavioral: Usual care — Subjects will continue with their usual healthcare routine and lifestyle. Upon completion of all study visits, subjects will be given access to the audio guides and information sheets for voluntary at-home practice exercises
  Arms: Usual care group

SUMMARY:
The goal of this study is to evaluate the feasibility and acceptability of a revised 4-week mindfulness program among young women with elevated stress and anxiety in Puerto Rico

DETAILED DESCRIPTION:
Women in Puerto Rico (PR) experience a high prevalence of cardiometabolic diseases (CMD), with 38% affected by obesity and 42% by hypertension. These rates are higher than those observed in PR men and non-Latinx White women in the continental U.S. Chronic stress is a key risk factor for CMD, and PR women report higher psychological distress than men, despite facing similar social and environmental stressors. Young adult women are particularly vulnerable, as stress during this life stage can shape long-term health outcomes, highlighting the need for targeted interventions.

Mindfulness-Based Stress Reduction (MBSR) is a structured, evidence-based program designed to reduce stress through techniques such as focused attention, open monitoring, and non-judgmental awareness. MBSR has been shown to lower blood pressure, improve heart rate variability (HRV), and reduce psychological distress, including anxiety and depression. The program's emphasis on group sessions aligns well with PR's collectivist culture, making it a potentially effective approach for this population. However, traditional MBSR programs, which span eight weeks with long session durations and extensive home practice, pose feasibility challenges, particularly in PR, where transportation and time constraints are significant barriers.

To overcome these limitations, researchers have adopted a 4-week MBSR program tailored specifically for young PR women, using shorter sessions and telehealth delivery. Preliminary research has demonstrated good participant retention, satisfaction, and improvements in psychological distress among Latinx women, but no randomized controlled trials (RCTs) have been conducted to evaluate MBSR's impact on PR women's cardiometabolic health. The proposed pilot RCT aims to address this gap by testing the feasibility, acceptability, and effectiveness of the adapted 4-week MBSR program, providing a culturally relevant intervention to reduce stress and improve CMD outcomes in this underserved group.

ELIGIBILITY:
Inclusion Criteria:

* Reporting female sex at birth
* Not identifying as a man, trans man, or trans woman.
* Individuals residing in Puerto Rico
* Spanish speaking
* Currently not pregnant
* Elevated stress (defined as a score >6 in the Perceived Stress Scale (PSS-4)34) or Elevated anxiety (defined as a score of 5 or more on the GAD-7 scale)
* Willing to undergo research activities.

Exclusion Criteria:

* Male sex at birth
* Identifying as a man, trans man, or trans woman.
* Currently pregnant
* Previous participation in an 8-week MBSR program
* Experiencing moderately severe or severe depressive symptoms (PHQ-9>15)35)
* Have active suicidal ideation (PHQ-9 item #9)35
* Self-report history of cognitive and psychiatric conditions
* Lack of access to the internet/phone (mode of focus group discussions-via Zoom)

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Not identifying as a man, trans man, or trans woman.
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rates of recruitment | Baseline
  Number of participants approached for the study versus number of participants that are enrolled.
Rates of retention | Baseline, 2 months follow up
  Number of participants at the beginning of the study versus the number of participants at the end of the study.
Rates of adherence | Post intervention (1-month), 2-month follow up
  Adherence will be measured by the number of phone sessions attended and the frequency of self-reported completed home practice, both assessed at post-intervention assessments.
Rates of satisfaction | Post intervention (1 month), 2 months follow up
  Ratings of satisfaction, also assessed by client satisfaction questionnaire (CSQ-8) in post-intervention assessments, will be measured with several questions, including one that reads "Overall, how satisfied were you with the stress reduction program", "How satisfied are you now (after the stress reduction program) with your ability to manage the stress in your life?", and "How much did the program helped you manage your stress?

SECONDARY OUTCOMES:
Change in Depression symptoms | Baseline, Post intervention (1 month), 2 months follow up
  Center for Epidemiological Studies Depression (CESD) 10-item scale, which asks about the frequency of depressed mood, guilt, worthlessness, helplessness, hopelessness, loss of appetite, and sleep disturbance. Score ranges from 0 to 30, with higher scores meaning more depressive symptoms.
Change in Anxiety (GAD-& score) | Baseline, Post intervention (1 month), 2 months follow up
  GAD-7 scale, which asks about the frequency of feeling nervous, unable to stop worrying, trouble relaxing, and being easily irritable.
  It includes 7 questions, each scored from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21. A score of 10 or more suggests clinically significant anxiety and may indicate the need for further evaluation.
Change in PTSD symptoms | Baseline, Post intervention (1 month), 2 months follow up
  Civilian Abbreviated Scale from the PTSD Checklist (PCL), which assesses repeated disturbing memories of a stressful past event.
  It typically includes 4 to 6 items, focusing on key symptom clusters from the DSM, such as: Intrusive thoughts (e.g., repeated, disturbing memories of a stressful event) Avoidance of reminders, Negative mood or thoughts, Hyperarousal (e.g., being easily startled)
  Each item is rated on a 5-point scale from "Not at all" to "Extremely". Higher scores indicate more severe symptoms and may suggest the need for further evaluation.
Change in perceived symptoms | Baseline, Post intervention (1 month), 2 months follow up
  Perceived Stress Scale (PSS-4) measures the degree to which someone perceives their life situations as overwhelming, uncontrollable, and unpredictable.
  4 items rated on a 5-point Likert scale (0 = Never to 4 = Very often). Higher scores mean greater perceived stress
Change in blood pressure | Baseline, Post intervention (1 month), 2 months follow up
  Systolic and diastolic blood pressure will be measured three times, in the sitting position (after a 5-min rest), using an electronic sphygmomanometer (OMRON). Measures will be averaged
Change in adiposity | Baseline, Post intervention (1 month), 2 months follow up
  BMI will be calculated from measured weight (light clothes) and height (no shoes).
  Waist circumference will be measured twice (cm) with a Gulick II Plus tape; measures will be averaged
Heart rate variability (HRV) | Baseline, Post intervention (1 month), 2 months follow up
  Fitbit Luxe is a device that measures HRV using the root mean square of successive differences equation72 and has been utilized to assess HRV in research studies. Participants will be instructed to wear the device daily throughout the study period. Data will be abstracted through the device's porta

CONTACTS AND LOCATIONS:
Overall Officials: Andrea López-Cepero, PhD, Principal Investigator — Rollins School of Public Health

IPD SHARING:
Plan to Share IPD: Yes
Data on the following variables may be shared: psychological distress (depression symptoms, anxiety symptoms, PTSD symptoms), resilience (shift and persist, mindfulness), health behaviors (smoking, eating habits), weight, blood pressure, height, sociodemographic (socioeconomic variables, age), number of sessions attended and practice exercise completed.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting January 2027